CLINICAL TRIAL: NCT00005710
Title: Recycling of Chronic Smokers to Sustained Abstinence
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4919; R01HL044992 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Lung Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Lung Diseases

SUMMARY:
To develop and to test a brief telephone intervention following clinic treatment for smoking cessation.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

A total of 1,083 chronic smokers were randomly assigned either to a traditional state-of-the-art smoking cessation clinic or to the clinic supplemented by telephone support for recycling. Telephone outreach consisted of three separate rounds of intervention three months, nine months, and 21 months after the targeted date for quitting in the smoking cessation clinics.

Telephone calls to abstinent subjects reinforced success and offered advice and support in coping with difficult situations. Calls to relapsers and nonabstainers debriefed concerning the relapse episode (as appropriate) and encouraged subjects to initiate concrete action toward quitting including setting a quit date. Subjects were offered self-help materials as well as referrals to more intensive programs.

Follow-up data collection was separate from recycling contacts and occured six, 12, 24, and 34 months after the initial smoking cessation clinics. Projected longterm sustained abstinence rates were 35 percent for recycling and 25 percent for the clinic only comparison. If results were as predicted, an effective low-cost telephone outreach protocol was made available that could dramatically assist in smoking cessation and thereby substantially reduce cardiovascular disease.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07; Study Completion 1995-06

REFERENCES:
- [Background] Roski J, Schmid LA, Lando HA. Long-term associations of helpful and harmful spousal behaviors with smoking cessation. Addict Behav. 1996 Mar-Apr;21(2):173-85. doi: 10.1016/0306-4603(95)00047-x. PMID 8730519
- [Background] Lando HA, Pirie PL, Roski J, McGovern PG, Schmid LA. Promoting abstinence among relapsed chronic smokers: the effect of telephone support. Am J Public Health. 1996 Dec;86(12):1786-90. doi: 10.2105/ajph.86.12.1786. PMID 9003138
- [Background] Lichtenstein E, Glasgow RE, Lando HA, Ossip-Klein DJ, Boles SM. Telephone counseling for smoking cessation: rationales and meta-analytic review of evidence. Health Educ Res. 1996 Jun;11(2):243-57. doi: 10.1093/her/11.2.243. PMID 10163409